CLINICAL TRIAL: NCT05329571
Title: Microbiome Correlates of Dietary Interventions in Patients With Fibromyalgia and Their Association With Symptom Modification
Brief Title: The Effects of Dietary Changes on Gut-bacteria and Fibromyalgia Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Louise and Alan Edwards Foundation (Unknown)
Responsible Party: Principal Investigator, Dr. Yoram Shir, Director of the Alan Edwards Pain Management Unit, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Diet-FM/2020-6134
Record Dates: First submitted 2022-02-22; First posted 2022-04-15 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Fibromyalgia; Diet, Gluten-Free
MeSH Terms: conditions — Fibromyalgia | interventions — FODMAP Diet; Diet, Gluten-Free; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-FODMAP Diet (Experimental): Participants will be instructed to maintain their usual diet, while eliminating FODMAPs (A subgroup of carbohydrates are considered fermentable, given the lack of suitable hydrolase enzymes in the colon, required for their digestion and absorption, thus making them available for fermentation).
  Interventions: Behavioral: Low-FODMAP diet
- Gluten-Free Diet (Experimental): Participants will be instructed to maintain their usual diet, while eliminating all dietary gluten.
  Interventions: Behavioral: Gluten-free Diet
- Control (Other): Patients of this group will be asked to adhere to their regular, daily diet.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Low-FODMAP diet — Participants will be instructed to maintain their usual diet, while eliminating all dietary gluten.
  Arms: Low-FODMAP Diet
Behavioral: Gluten-free Diet — Participants will be instructed to maintain their usual diet, while eliminating all dietary gluten.
  Arms: Gluten-Free Diet
Behavioral: Control group — Patients of this group will have dietary consultation but will not change their regular diet for the period of the study.
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the efficacy of two diets - gluten-free and low-FODMAP diet- in relieving symptoms of fibromyalgia, and study whether these changes could be associated with changes in the gut microbiome (gut bacteria).

ELIGIBILITY:
Inclusion Criteria:

1. Women over the age of 18, diagnosed with FM.
2. Chronic widespread pain index >= 9 and pain intensity >= 6.
3. Able to read and write in either French or English.

Exclusion Criteria:

1. Any major illness (e.g. malignancy, active inflammatory disease, metabolic disease, etc.)
2. Inflammatory bowel disease.
3. Severe depression (HADS score for depression > 10).
4. Current use of LFD or GFD.
5. Pregnancy
6. Vegan diet

The inclusion/exclusion criteria were set to reduce the risk of confounding factors that could affect gut microbiota composition. To date, information on microbiome alterations in individuals with fibromyalgia is only available for female patients, and thus recruitment will be limited to women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-03-12 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in gut microbiome composition in response to dietary intervention | Four weeks after the initiation of the new diet compared to baseline.
  Genome structure, structural variants - Differential abundance analysis will be performed using 16S rRNA.
Changes in stool microbiota-related metabolites affecting host physiology, in response to dietary intervention. | Four weeks after the initiation of the new diet compared to baseline.
  Metabolomics analysis will be performed (Metabolon, USA) - targeted metabolomic for bile acids and SCFA analysis.
Changes in blood microbiota-related metabolites, affecting host physiology, in response to dietary intervention | Four weeks after the initiation of the new diet compared to baseline.
  Metabolomics analysis will be performed (Metabolon, USA) - targeted metabolomic for bile acids and SCFA analysis.

SECONDARY OUTCOMES:
The Fibromyalgia Survey Diagnostic Criteria and Severity Scale (FSDC) scores. | Four weeks after the initiation of the new diet compared to baseline.
  assessing symptom severity, pain distribution, fatigue, sleep quality and cognitive and somatic complaints in fibromyalgia patients.
  A questionnaire assessing symptom severity, pain distribution, fatigue, sleep quality and cognitive and somatic complaints in fibromyalgia patients.
The Fibromyalgia Impact Questionnaire (FIQ) score | Four weeks after the initiation of the new diet compared to baseline.
  A 10 items questionnaire evaluating physical functioning, work difficulty, pain, fatigue, morning tiredness, stiffness, anxiety and depression.
Hospital Anxiety and Depression Scale (HADS) score | Four weeks after the initiation of the new diet compared to baseline.
  A 14-items questionnaire assessing the level of depression and anxiety.
The Pittsburg Sleep Quality Index scores | Four weeks after the initiation of the new diet compared to baseline.
  An 11 item sleep quality evaluation questionnaire.
ROME IV criteria for irritable bowel syndrome | Four weeks after the initiation of the new diet compared to baseline.
  Four yes-or-no items

CONTACTS AND LOCATIONS:
Overall Officials: Yoram Shir, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Alan Edwards Pain Management Unit - Montreal General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bauer KC, Huus KE, Finlay BB. Microbes and the mind: emerging hallmarks of the gut microbiota-brain axis. Cell Microbiol. 2016 May;18(5):632-44. doi: 10.1111/cmi.12585. Epub 2016 Mar 31. PMID 26918908
- [Background] Minerbi A, Gonzalez E, Brereton NJB, Anjarkouchian A, Dewar K, Fitzcharles MA, Chevalier S, Shir Y. Altered microbiome composition in individuals with fibromyalgia. Pain. 2019 Nov;160(11):2589-2602. doi: 10.1097/j.pain.0000000000001640. PMID 31219947
- [Background] Thaiss CA, Itav S, Rothschild D, Meijer MT, Levy M, Moresi C, Dohnalova L, Braverman S, Rozin S, Malitsky S, Dori-Bachash M, Kuperman Y, Biton I, Gertler A, Harmelin A, Shapiro H, Halpern Z, Aharoni A, Segal E, Elinav E. Persistent microbiome alterations modulate the rate of post-dieting weight regain. Nature. 2016 Dec 22;540(7634):544-551. doi: 10.1038/nature20796. Epub 2016 Nov 24. PMID 27906159
- [Background] Tong M, Li X, Wegener Parfrey L, Roth B, Ippoliti A, Wei B, Borneman J, McGovern DP, Frank DN, Li E, Horvath S, Knight R, Braun J. A modular organization of the human intestinal mucosal microbiota and its association with inflammatory bowel disease. PLoS One. 2013 Nov 19;8(11):e80702. doi: 10.1371/journal.pone.0080702. eCollection 2013. PMID 24260458
- [Background] Zhang X, Zhang D, Jia H, Feng Q, Wang D, Liang D, Wu X, Li J, Tang L, Li Y, Lan Z, Chen B, Li Y, Zhong H, Xie H, Jie Z, Chen W, Tang S, Xu X, Wang X, Cai X, Liu S, Xia Y, Li J, Qiao X, Al-Aama JY, Chen H, Wang L, Wu QJ, Zhang F, Zheng W, Li Y, Zhang M, Luo G, Xue W, Xiao L, Li J, Chen W, Xu X, Yin Y, Yang H, Wang J, Kristiansen K, Liu L, Li T, Huang Q, Li Y, Wang J. The oral and gut microbiomes are perturbed in rheumatoid arthritis and partly normalized after treatment. Nat Med. 2015 Aug;21(8):895-905. doi: 10.1038/nm.3914. Epub 2015 Jul 27. PMID 26214836
- [Background] Lowry E, Marley J, McVeigh JG, McSorley E, Allsopp P, Kerr D. Dietary Interventions in the Management of Fibromyalgia: A Systematic Review and Best-Evidence Synthesis. Nutrients. 2020 Aug 31;12(9):2664. doi: 10.3390/nu12092664. PMID 32878326